CLINICAL TRIAL: NCT00768729
Title: Immunosuppression Minimization to Single Drug Therapy With Sirolimus (Rapamune) in Pediatric Transplantation
Brief Title: Safety of Immunosuppression Minimization in Children and Adolescents After Kidney Transplantation
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: DAIT CTOTC-01
Record Dates: First submitted 2008-10-06; First posted 2008-10-08 (Estimated); Last update posted 2013-02-15 (Estimated); Status verified 2013-02

CONDITIONS: Kidney Failure, Chronic; Kidney Transplantation; Immunosuppression
Keywords: End stage renal disease; Kidney transplantation; Renal transplantation; Kidney failure; Children; Adolescents; Sirolimus; Rapamycin; CellCept; Mycophenolate mofetil (MMF); Azathioprine
MeSH Terms: conditions — Kidney Failure, Chronic; Renal Insufficiency | interventions — Sirolimus; Azathioprine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental): Participants who have been maintained on MMF at study entry will start the study on 600 mg/m2 MMF orally daily. Participants who have been maintained on Azathioprine due to MMF intolerance will receive 1 mg/kg Azathioprine orally daily.
  Participants will continue receiving sirolimus throughout the study. However, MMF or Azathioprine will be withdrawn gradually over a period of at least 6 months. Dosage will be reduced by 25% initially and by 25% every subsequent 2 months resulting in complete withdrawal by 6 months.
  Interventions: Drug: Sirolimus; Drug: MMF or Azathioprine

INTERVENTIONS:
Drug: Sirolimus — Oral tablets or liquid taken every 12 hours. Dosage adjusted to attain target trough levels of 8-12 ng/mL. Participants who have maintained such levels at study entry on once daily dosage will be permitted to continue on once daily dosing.
  Other Names: Rapamycin, Rapamune
Drug: MMF or Azathioprine — 600 mg/m2 MMF taken orally daily or Azathioprine orally daily. Dosage of Azathioprine is dependent on weight. MMF or Azathioprine will be reduced by 25% initially and by 25% every 2 months resulting in complete withdrawal by 6 months.

SUMMARY:
Kidney transplantation is widely considered to be the treatment of choice for children with End Stage Renal Disease (ESRD). The purpose of this study is to determine the safety of sirolimus monotherapy for long-term immunosuppression in children and adolescents after kidney transplantation.

DETAILED DESCRIPTION:
Improvements in surgical techniques, donor selection, immunosuppression practices, and the enhanced experience of specialized pediatric transplant teams have all led to marked improvements in patient and kidney graft survival in infants and young children Long-term graft survival rates decrease in adolescents 11 to 17 years of age. Several studies have suggested this decrease may be the result of noncompliance with immunosuppressive medications in this age group. Therefore, protocols that minimize the use of immunosuppressive medications, while retaining kidney function are necessary for improving graft and patient survival in children. The purpose of this study is to determine the safety of sirolimus monotherapy for long-term immunosuppression in children and adolescents after kidney transplantation.

This study will enroll 10 participants who previously completed the CCTPT-PC01 study. The accrual period is scheduled for 12 months. The study follow-up period will last 96 weeks. Patients from the CCTPT-PC01 study have been maintained on sirolimus and mycophenolate mofetil (MMF) since 2-3 months post transplant. Enrolled participants receiving (MMF) or Azathioprine at study entry will have their doses withdrawn gradually over a period of 6 months. Dosage will be reduced by 25% initially and by 25% every 2 months resulting in complete withdrawal by 6 months.

This study will consist of 11 study visits after screening and study entry. Study visits will occur at weeks 1, 8, 16, 24, 32, 40, 48, 60, 72, 84, and 96. A physical exam, vital signs, sirolimus levels, as well as blood and urine collection will occur at all visits. A renal biopsy will be performed at week 96.

ELIGIBILITY:
Inclusion Criteria:

* Participant and/or parent guardian able to understand and willing to provide informed consent
* Previously enrolled and completed the CCTPT-PC01 study and within the 36 months post-completion timeframe prior to study entry
* Currently receiving sirolimus and MMF or azathioprine therapy
* No history of acute rejection episodes
* No evidence of acute or chronic rejection on the 24 month CCTPT-PC01 protocol biopsy or any subsequent biopsy obtained after that time prior to study entry
* PRA (Class I and II) less than 5% at study entry
* No evidence of donor specific antibody at study entry
* Stable renal function with GFR greater than 60 cc/min 1.73M^2 using the Schwartz calculated method
* A negative pregnancy test for female participants of childbearing potential at study entry
* Agreement by female and male participants to use FDA approved methods of contraception.

Exclusion Criteria:

* Total lymphocyte count less than 400 mm^3
* Acute or chronic infection at study entry
* Treatment with investigational drug within 1 month prior to study entry
* Mental illness or history of drug or alcohol abuse that, in the opinion of the investigator, would interfere with the study
* History of allergic reaction to Iodine GFR assay
* History of malignancy within the past 12 months
* Inability or unwillingness to give informed consent or comply with the study protocol

Ages: 1 Year to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 7 (Actual)
Dates: Start 2009-05; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Per-person incidence of acute rejection episodes and death or graft loss | Throughout study

SECONDARY OUTCOMES:
Incidence of chronic allograft dysfunction | Throughout study
Incidence of sub-clinical rejection | Throughout study
Incidence of hospitalizations | Throughout study
Incidence of surgical complications | Throughout study
Resumption of MMF or other therapy | Throughout study
Incidence, severity, and treatment of anemia, hypertension, hyperlipidemia, proteinuria, thrombocytopenia, and leukopenia | Throughout study
Incidence, severity, and treatment of opportunistic infections | Throughout study
Incidence of biopsy proven PTLD | Throughout study
Renal function assessed by measured GFR | At baseline, week 48 and week 96
Development of donor-specific or non-specific anti-HLA antibodies | Throughout study
Evolution of immune response in cellular, humoral, and molecular assays from baseline through week 96 | Throughout study

CONTACTS AND LOCATIONS:
Overall Officials: William H. Harmon, MD, Study Chair — Boston Children's Hospital
Locations (5):
- United States (5):
  - Children's Hospital of Central California, Madera, California
  - UCSF Children's Hospital, San Francisco, California
  - Children's Hospital, Boston, Boston, Massachusetts
  - Children's Hospital, Philadelphia, Philadelphia, Pennsylvania
  - Children's Hospital and Regional Medical Center, Seattle, Seattle, Washington

REFERENCES:
- [Background] McDonald RA, Smith JM, Ho M, Lindblad R, Ikle D, Grimm P, Wyatt R, Arar M, Liereman D, Bridges N, Harmon W; CCTPT Study Group. Incidence of PTLD in pediatric renal transplant recipients receiving basiliximab, calcineurin inhibitor, sirolimus and steroids. Am J Transplant. 2008 May;8(5):984-9. doi: 10.1111/j.1600-6143.2008.02167.x. PMID 18416737
- [Background] Watson CJ, Bradley JA, Friend PJ, Firth J, Taylor CJ, Bradley JR, Smith KG, Thiru S, Jamieson NV, Hale G, Waldmann H, Calne R. Alemtuzumab (CAMPATH 1H) induction therapy in cadaveric kidney transplantation--efficacy and safety at five years. Am J Transplant. 2005 Jun;5(6):1347-53. doi: 10.1111/j.1600-6143.2005.00822.x. PMID 15888040
- See also: CTOTC Website — https://www.ctotc.org